CLINICAL TRIAL: NCT03272022
Title: Micronutrient Status in Pregnant and Lactating Women and Their Infants
Brief Title: Micronutrient Status During Pregnancy
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/2447
Record Dates: First submitted 2017-08-30; First posted 2017-09-05 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Deficiency Vitamins
Keywords: cobalamin, folate
MeSH Terms: conditions — Avitaminosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma from never-pregnant, pregnant and lactating women and infants aged six months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women: never-pregnant women
- pregnant women: pregnant

SUMMARY:
An adequate micronutrient status during fetal life and infancy is important for optimal development. Dietary practices during pregnancy, lactation and infancy vary among populations and there is today no clear agreement on what constitutes the best diet, including micronutrient supplementation, during this period. There is consequently no clear agreement on what constitutes an optimal biochemical micronutrient status in mothers and infants. Due to substantial physiological changes in plasma volume, hormones, transport proteins and organ function during these periods, the ordinary reference levels or cut off levels used for biochemical assessment of micronutrient status are unsuited to these groups of patients.

The objective of the study is to establish cut off levels for important vitamins and trace elements during pregnancy, lactation and infancy in order to ensure an optimal infant neurodevelopment and to study how micronutrient status influence the immunosystem.

DETAILED DESCRIPTION:
The investigators have analyzed micronutrients, including all vitamins and trace elements and related aminoacids and markers of cellular immunoactivation in 160 fertile, unpregnant women, 115 pregnant women from pregnancy week 18, throughout pregnancy and the first 6 postpartum months and their infant at 6 months. Infant gross motor development is associated with micronutrient status, so the investigators will relate gross motor development at 6 months to maternal micronutrient status during pregnancy and postpartum, in order to establish relevant cut off levels for micronutrients and related biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* healthy never-pregnant and pregnant women

Exclusion Criteria:

chronic illness-

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — pregnant women and never-pregnant women
Study Population: healthy never-pregnant (n =158) and pregnant women (n=114) and their infants (n=114)
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2011-12-14 (Actual); Primary Completion 2016-02-08 (Actual); Study Completion 2016-02-08 (Actual)

PRIMARY OUTCOMES:
Change in micronutrient status during pregnancy and lactation | The investigators will study change in micronutrients during pregnancy and lactation
  Determine adequate vitamin levels in pregnancy and lactation

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Mellgren, MD, PhD, Study Director — Haukeland University Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Green R, Allen LH, Bjorke-Monsen AL, Brito A, Gueant JL, Miller JW, Molloy AM, Nexo E, Stabler S, Toh BH, Ueland PM, Yajnik C. Vitamin B12 deficiency. Nat Rev Dis Primers. 2017 Jun 29;3:17040. doi: 10.1038/nrdp.2017.40. PMID 28660890
- [Result] Torsvik IK, Ueland PM, Markestad T, Midttun O, Bjorke Monsen AL. Motor development related to duration of exclusive breastfeeding, B vitamin status and B12 supplementation in infants with a birth weight between 2000-3000 g, results from a randomized intervention trial. BMC Pediatr. 2015 Dec 18;15:218. doi: 10.1186/s12887-015-0533-2. PMID 26678525
- [Result] Torsvik I, Ueland PM, Markestad T, Bjorke-Monsen AL. Cobalamin supplementation improves motor development and regurgitations in infants: results from a randomized intervention study. Am J Clin Nutr. 2013 Nov;98(5):1233-40. doi: 10.3945/ajcn.113.061549. Epub 2013 Sep 11. PMID 24025626
- [Result] Bjorke-Monsen AL, Torsvik I, Saetran H, Markestad T, Ueland PM. Common metabolic profile in infants indicating impaired cobalamin status responds to cobalamin supplementation. Pediatrics. 2008 Jul;122(1):83-91. doi: 10.1542/peds.2007-2716. PMID 18595990
- [Result] Bjorke Monsen AL, Ueland PM, Vollset SE, Guttormsen AB, Markestad T, Solheim E, Refsum H. Determinants of cobalamin status in newborns. Pediatrics. 2001 Sep;108(3):624-30. doi: 10.1542/peds.108.3.624. PMID 11533328
- [Derived] Bjorke-Monsen AL, Varsi K, Averina M, Brox J, Huber S. Perfluoroalkyl substances (PFASs) and mercury in never-pregnant women of fertile age: association with fish consumption and unfavorable lipid profile. BMJ Nutr Prev Health. 2020 Nov 4;3(2):277-284. doi: 10.1136/bmjnph-2020-000131. eCollection 2020 Dec. PMID 33521539
- [Derived] Varsi K, Ueland PM, Torsvik IK, Bjorke-Monsen AL. Maternal Serum Cobalamin at 18 Weeks of Pregnancy Predicts Infant Cobalamin Status at 6 Months-A Prospective, Observational Study. J Nutr. 2018 May 1;148(5):738-745. doi: 10.1093/jn/nxy028. PMID 29947806